CLINICAL TRIAL: NCT07401446
Title: Comparison of Complication Rates of Onlay vs Sublay Mesh Repair of Incisional Hernia
Brief Title: Complication Rate of Onlay vs Sublay Mesh Repair in Incisional Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Gohar Ali, Principal Investigator, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMC-QAD-F No. IREB-1221
Record Dates: First submitted 2026-01-16; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Hernia; Ventral Hernia Repair; Incisional Hernia Repair; Abdominal Wall Hernia; Synthetic Mesh
Keywords: incisional Hernia; Mesh repair; Onlay Mesh repair; sublay Mesh Repair
MeSH Terms: conditions — Hernia; Hernia, Abdominal; Incisional Hernia

STUDY DESIGN:
Intervention Model Description: This study uses a parallel group randomized design in which eligible participants were randomly assigned to one of two intervention arms. One group underwent sublay mesh repair, and the other group underwent onlay mesh repair for incisional hernia. Participants received only the intervention assigned to their group, and outcomes were compared between the two groups over a three-month follow-up period.
Masking Description: This was an open-label study. Due to the nature of the surgical interventions, neither participants nor healthcare providers nor outcome assessors were blinded to the assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublay Mesh Repair (Experimental): Patients underwent open incisional hernia repair with placement of polypropylene mesh in the retromuscular preperitoneal (sublay) plane.
  Interventions: Procedure: Sublay Mesh Repair
- Onlay Mesh Repair (Active Comparator): Patients underwent open incisional hernia repair with placement of polypropylene mesh over the anterior rectus sheath (onlay technique).
  Interventions: Procedure: Onlay Mesh Repair

INTERVENTIONS:
Procedure: Sublay Mesh Repair — Patients underwent open incisional hernia repair with placement of polypropylene mesh in the retromuscular preperitoneal (sublay) plane.
  Arms: Sublay Mesh Repair
Procedure: Onlay Mesh Repair — Placement of polypropylene mesh over the anterior rectus sheath during open incisional hernia repair.
  Arms: Onlay Mesh Repair

SUMMARY:
This randomized controlled trial was conducted at the Department of Surgery, Hayatabad Medical Complex, Peshawar. Eligible patients with incisional hernia were randomized into two parallel groups: sublay mesh repair and onlay mesh repair. Procedures were performed by a single experienced general surgeon. Postoperative complications were assessed by an independent surgeon blinded to the type of procedure. Patients were followed for a period of three months to evaluate safety and recurrence outcomes.

DETAILED DESCRIPTION:
Incisional hernia is a frequent postoperative complication following abdominal surgery and represents a significant source of morbidity due to discomfort, impaired quality of life, and risk of recurrence. Mesh reinforcement has become the standard approach for incisional hernia repair; however, the optimal anatomical position of mesh placement remains debated. Among the commonly used techniques, onlay mesh repair involves placement of mesh over the anterior rectus sheath, while sublay mesh repair places the mesh in the retromuscular preperitoneal plane. Each technique differs in operative dissection, tissue handling, and potential risk of postoperative complications.

This randomized controlled trial was conducted at the Department of Surgery, Hayatabad Medical Complex, Peshawar, to compare postoperative outcomes of onlay versus sublay mesh repair in patients undergoing elective incisional hernia repair. Adult patients aged 18 to 60 years presenting with incisional hernia and meeting predefined eligibility criteria were enrolled after providing written informed consent. Patients with recurrent, strangulated, or obstructed hernias, severe comorbid conditions, high anesthetic risk, or morbid obesity were excluded to minimize confounding factors.

Eligible participants were randomly allocated into two parallel groups using a lottery method. Patients assigned to Group A underwent sublay mesh repair, while those in Group B received onlay mesh repair. All surgical procedures were performed by a single experienced general surgeon to ensure procedural consistency. Standardized perioperative care protocols were followed for all patients.

Postoperatively, patients were monitored during hospital admission and followed in outpatient clinics for a period of three months. Assessment of postoperative complications, including wound infection, seroma, hematoma, and hernia recurrence, was carried out by an independent surgeon who was blinded to the surgical technique used. This masking approach was adopted to reduce assessment bias.

The primary objective of the study was to compare the overall postoperative complication rates between the two mesh placement techniques. Secondary objectives included evaluation of individual complication rates and recurrence during the follow-up period. Data were collected using a structured proforma and analyzed using standard statistical methods to determine differences between groups.

The findings of this study aim to provide evidence-based guidance regarding the safety and effectiveness of mesh placement techniques in incisional hernia repair and to assist surgeons in selecting an optimal approach that minimizes postoperative complications and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Patients diagnosed with primary incisional hernia on clinical examination.
* Hernia suitable for open surgical repair with mesh.
* Both male and female patients.
* Patients able and willing to provide written informed consent.

Exclusion Criteria:

* Obstructed or strangulated hernia on presentation.
* Recurrent incisional hernia.
* Patients with BMI > 40.
* Patients with debilitating chronic diseases, including:
* Chronic liver disease
* Chronic renal impairment
* Chronic cardiac disease
* Chronic pulmonary disease
* Patients with American Society of Anesthesiologists (ASA) physical status ≥ 3.
* Patients unfit for general anesthesia.
* Patients unable or unwilling to follow up for postoperative assessment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Complication Rate | 30 days after surgery
  Incidence of complications within 30 days after surgery, including wound infection, seroma, hematoma, and hernia recurrence, in patients undergoing onlay versus sublay mesh repair of incisional hernia.

SECONDARY OUTCOMES:
Length of Hospital Stay | Number of days From enrollment up to the hospital discharge
  Duration of hospitalization following surgery in both study groups for this single disease.
Hernia Recurrence Rate | Assessed at 6 months and 12 months after surgery
  Number of patients with hernia recurrence within 6 months and 12 months postoperatively.
Operative Time | During the index surgical procedure (from skin incision to skin closure)
  Total duration of surgery from incision to closure for onlay and sublay procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) from this study has not yet been finalized. Considerations regarding patient privacy, data de-identification, and institutional policies on data sharing are still under review. Once these factors are addressed, a detailed plan for data sharing may be developed in compliance with ethical guidelines and institutional requirements.

REFERENCES:
- [Result] Burger JW, Luijendijk RW, Hop WC, Halm JA, Verdaasdonk EG, Jeekel J. Long-term follow-up of a randomized controlled trial of suture versus mesh repair of incisional hernia. Ann Surg. 2004 Oct;240(4):578-83; discussion 583-5. doi: 10.1097/01.sla.0000141193.08524.e7. PMID 15383785
- [Result] Walming S, Angenete E, Block M, Bock D, Gessler B, Haglind E. Retrospective review of risk factors for surgical wound dehiscence and incisional hernia. BMC Surg. 2017 Feb 22;17(1):19. doi: 10.1186/s12893-017-0207-0. PMID 28222776
- [Result] Pereira C, Gururaj S. Onlay Versus Sublay Mesh Repair for Incisional Hernias: A Systematic Review. Cureus. 2023 Jan 24;15(1):e34156. doi: 10.7759/cureus.34156. eCollection 2023 Jan. PMID 36713818
- [Result] Kohler A, Beldi G. [Recurrence after hernia surgery: complication or natural course?] Chirurg. 2014 Feb;85(2):112-6.
- [Result] Rayman S, Gorgov E, Assaf D, Carmeli I, Nevo N, Rachmuth J, Mnouskin Y. Quality of life, post-operative complications, and hernia recurrence following enhanced-view Totally Extra-Peritoneal (eTEP) Rives-Stoppa for incisional and primary ventral hernia repair. Updates Surg. 2023 Oct;75(7):1971-1978. doi: 10.1007/s13304-023-01572-x. Epub 2023 Jun 28. PMID 37378814
- [Result] Omar I, Zaimis T, Townsend A, Ismaiel M, Wilson J, Magee C. Incisional Hernia: A Surgical Complication or Medical Disease? Cureus. 2023 Dec 15;15(12):e50568. doi: 10.7759/cureus.50568. eCollection 2023 Dec. PMID 38222215

DOCUMENTS (2):
  • Study Protocol (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07401446/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07401446/SAP_001.pdf